CLINICAL TRIAL: NCT06875154
Title: Influence of Original Native Tricuspid Valve Lesion (Stenosis or Steno-insufficiency or Insufficiency) on Post-implant Structural Bioprosthetic Degeneration After Tricuspid Valve Replacement.
Acronym: DURABLE-TRIC
Status: Enrolling by invitation | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Roberto Lorusso, Prof. MD PhD, Maastricht University Medical Center
Other Study IDs: 2023-0324
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Degeneration of Tricuspid Surgical Bioprosthesis
Keywords: tricuspid valve; Tricuspid bioprosthesis; Durability
MeSH Terms: interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Surgical Tricuspid bioprosthesis: All patients undergoing elective tricuspid valve replacement from 2000 to 2020. All operations were performed through median longitudinal sternotomy, mini-sternotomy or mini- thoracotomy.Intraoperative transesophageal echocardiography (TOE) was used in all patients. Arterial cannulation was central and venous cannulation was achieved with a common two-stage cannula in the right atrium. Left ventricle was vented through the right superior pulmonary vein.In minimally invasive procedures, venous cannulation was achieved percutaneously. Myocardial protection was achieved by administration of cold crystalloid or blood cardioplegia at the surgeon's discretion in an antegrade (indirect or selective) or retrograde fashion.
  Beating heart procedure can be performed without the use of aortic clamp. The prosthesis were be implanted with 2-0 U-shaped sutures.
  Interventions: Procedure: Valve replacement

INTERVENTIONS:
Procedure: Valve replacement — All operations were performed through median longitudinal sternotomy or mini-sternotomy or minitoracothomy Intraoperative transesophageal echocardiography (TOE) was used in all patients. Arterial cannulation was central and venous cannulation was achieved with a common two-stage cannula in the right atrium or from peripheral access. Left ventricle was vented through the right superior pulmonary vein.
  In minimally invasive procedures, venous cannulation was achieved percutaneously. Myocardial protection was achieved by administration of cold crystalloid or blood cardioplegia at the surgeon's discretion in an antegrade (indirect or selective) or retrograde fashion.. All the prosthesis were be implanted with supranular technique and 2-0 U-shaped pledgeted sutures.

SUMMARY:
The structural deterioration process of the implanted bioprosthesis in tricuspid position for tricuspid valve pathology is gradual and irreversible and includes many changes, such as pannus growth, leaflet fibrosis and calcification, delamination of the connective tissue, ruptures and perforations of leaflets. In the great majority of cases SVD consists of leaflet calcium deposits and can be clinically associated with young age, hypercholesterolemia, hypertension, diabetes mellitus, renal failure. The long term durability of these bioprosthesis is still missing.

DETAILED DESCRIPTION:
It is not clear if the same biochemical, hemodynamic and immunological mechanisms leading to native valve calcification can cause bioprosthetic SVD. We hypothesize that the mechanisms protecting the native valve from calcification in the insufficiency disease may subsequently protect also the bioprosthetic valve from calcific SVD. In such a case, considering also the reduced incidence in insufficiency patients of prosthesis-patient mismatch, supposedly associated with increased risk of SVD, indication for bioprosthetic valve use could be expanded in patients with insufficiency. Because of the rising demand of bioprosthetic valve implantation, even a few years increase in the expected durability of the BHV, although limited to a defined population of patients, will have a very relevant clinical impact.

We aim to perform a retrospective, multi-center, observational study. All patients undergoing elective tricuspid valve replacement from 2000 to 2020 who met the inclusion criteria for the study (described in the dedicated section) will be enrolled in the study. These patients will be followed-up as part of routine care, and information about the clinical status, NYHA functional class, possible rehospitalization, possible cardiovascular events and postoperative echocardiography will be available for analysis. Once consent is given, and if required by local governance, pre-, intra- and post-operative data will be collected in a dedicated, structured, database.

ELIGIBILITY:
Inclusion Criteria:

- Age ≥ 18 years; 6

- Patients who underwent isolated tricuspid valve replacement for stenosis, regurgitation or steno-regurgitation

- Signed informed consent, inclusive of release of medical information where required by local governance.

Exclusion Criteria:

* Tricuspid valve replacement associated with other surgical procedures (CABG or other)

Previous cardiac surgery of any kind;

- Surgery for acute endocarditis

- Participation in another clinical trial that could interfere with the endpoints of this study.

- Pregnant or breastfeeding at time of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing elective tricuspid valve replacement from 2000 to 2020 who met the inclusion criteria for the study (described in the dedicated section) will be enrolled in the study
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Long term durability | 20 years
  Long term durability of the tricuspid bioprosthesis in terms of structural valve deterioration or /and associated complications.
  Echocardiographic parameters will be used. Continous variables will be implied.

SECONDARY OUTCOMES:
Long term survival | 20 years
  Long term survival, event free survival, freedom from reoperations and hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardio-Thoracic Surgery Department - Heart & Vascular Centre - Maastricht University Medical Centre (MUMC+), Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided